CLINICAL TRIAL: NCT05227066
Title: Efficacy of Adding Lower Extremity Weights on Balance in Children With Ataxic Cerebral Palsy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, walaa eldesoukey heneidy, lecturer of physical therapy, Delta University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ataxic CP
Record Dates: First submitted 2022-01-06; First posted 2022-02-07 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2024-12

CONDITIONS: Ataxic Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy, Ataxic, Autosomal Recessive

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional physical therapy group (Experimental): received traditional physical therapy protocol
  Interventions: Other: traditional physical therapy group
- lower extremity weights group (Experimental): received the same traditional physical therapy in addition to lower extremity weights
  Interventions: Other: adding lower extremity weights; Other: traditional physical therapy group

INTERVENTIONS:
Other: adding lower extremity weights — All children in the two groups received physical therapy protocol for 30 minutes in addition to half kg of sandbags weights attached for each leg
  Arms: lower extremity weights group
Other: traditional physical therapy group — traditional physical therapy group

SUMMARY:
Ataxic CP is one type of cerebral palsy. children with ataxic cerebral palsy have trouble with balance and coordination. They may walk with their legs farther apart than other kids and have a hard time with activities that use small hand movements, like writing. Some also have trouble with depth perception This means being able to accurately judge how close or far away something is

ELIGIBILITY:
Inclusion Criteria:

* ataxic cerebral palsy aged 7-13 years

Exclusion Criteria:

* any musculoskeletal conditions that affect balance previous surgeries that affecting balance

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2025-01-05 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Change in overall stability index | baseline and after 3 months of intervention.
  change in overall stability index will measured by using biodex balance system

SECONDARY OUTCOMES:
antero-posterior stability index | baseline and after 3 months of intervention.
  change in antero-posterior stability index will measured by using biodex balance system
mediolateral stability index | baseline and after 3 months of intervention.
  change in mediolateral stability index will measured by using biodex balance system

CONTACTS AND LOCATIONS:
Overall Officials: Hala I. Kassem, Professor, Study Director — Professor of physical therapy
Locations (1):
- Delta University for Science and Technology, Gamasa, Dakahelia, Egypt

IPD SHARING:
Plan to Share IPD: Yes